CLINICAL TRIAL: NCT00234741
Title: A Randomized, Double-Blind, Pilot Study of the Oral IL-12/23 Inhibitor, STA-5326 Mesylate, to Investigate Peripheral Blood and Mucosal Mononuclear Cell Phenotype and Cytokine Responses in Patients With Crohn's Disease
Brief Title: Study of STA-5326 Mesylate in Patients With Moderate to Severe Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Synta Pharmaceuticals Corp. (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 5326-11
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2008-12-04 (Estimated); Status verified 2008-12

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — apilimod

INTERVENTIONS:
Drug: STA-5326 mesylate

SUMMARY:
STA-5326 is an oral experimental drug that has been shown to block the release of interleukin-12 from peripheral blood mononuclear cells. Given this activity on the immune system, STA-5326 mesylate is a potential treatment for various autoimmune diseases, such as Crohn's disease, that are mediated by the inappropriate expression of Th1 cytokines.

This study is evaluating the use of STA-5326 mesylate in patients with moderate to severe, active Crohn's disease. Study visits include a screening visit, 4 treatment period visits over 4 weeks and a follow-up visit that will occur 7 days following the end of treatment. Subjects may continue treatment for an additional 4 weeks of open label STA-5326 mesylate administration that includes an additional 2 treatment period visits. Subjects will undergo a colonoscopy with biopsy collection at baseline, at the end of the 4 week blinded phase and at the end of the 4 week open label phase.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female aged 18 through 75 years.
* Has Crohn's disease diagnosed definitively prior to Screening (based upon clinical, endoscopic, radiologic imaging, or histological assessments).
* Has a CDAI score of 220 to 450, inclusive at Baseline.

Exclusion Criteria:

* Has any clinically significant disease (eg, renal, hepatic, neurological, cardiovascular, pulmonary, endocrinologic, psychiatric, hematologic, urologic, or other acute or chronic illness) that in the opinion of the investigator would make the subject an unsuitable candidate for this study.
* Is a woman who has a positive pregnancy test, who is breast-feeding, or who is sexually active without using birth control during the course of the study and Follow-up period.
* Is a woman of childbearing potential or a man who does not agree to use 2 forms of contraception during the course of the study and Follow-up period.
* Has clinically significant hematologic, hepatic or renal laboratory abnormalities.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2005-11

PRIMARY OUTCOMES:
To measure the changes from predose in peripheral blood and mucosal cytokines in subjects with active CD after administration of STA-5326 mesylate or placebo for 4 weeks

SECONDARY OUTCOMES:
To measure changes in other immunologic parameters.
To explore the level of cell-surface markers and specific gene expression patterns.
To measure changes in laboratory surrogate efficacy markers.
To measure the proportion of subjects in clinical remission at Day 29.
To measure the proportion of subjects with a clinical response at Day 29.
To measure the proportion of subjects with both clinical remission and clinical response at Day 29.
To confirm STA-5326 mesylate (and metabolite) levels in blood following oral administration to CD patients.
To measure the changes in endoscopic scores from Baseline to Day 29.
To measure the changes in the Inflammatory Bowel Disease Questionnaire overall score from Baseline to Day 29.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Mannon, MD, Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Nih/Niaid, Bethesda, Maryland, United States